CLINICAL TRIAL: NCT05289752
Title: Direct Versus Indirect Pick up of the Locator Retentive Caps for Two Implant-retained Mandibular Overdenture: Calibration of the Manufacturer Retentive Force and the Clinical Retention (Within-patient Study)
Brief Title: Direct Versus Indirect Pick up of the Locator Retentive Caps:(Within-patient Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A17030821
Record Dates: First submitted 2022-02-27; First posted 2022-03-21 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-02

CONDITIONS: Prosthesis Durability
MeSH Terms: conditions — Prosthesis Failure | interventions — Dental Implants; Denture, Overlay

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): GroupI: The retentive caps will be picked up by the indirect method on the cast first, then by the direct method.
  Interventions: Procedure: dental implants in the mandible; Device: locator attachment and overdenture
- Group II (Active Comparator): GroupII: The retentive caps will be picked up by the direct method on the cast first, then by the indirect method.
  Interventions: Procedure: dental implants in the mandible; Device: locator attachment and overdenture

INTERVENTIONS:
Procedure: dental implants in the mandible — placement of two interforaminal dental implants in the canine region in the mandible
Device: locator attachment and overdenture — placement of locator attachment and insertion of mandibular overdenture

SUMMARY:
The purpose of this study will be to evaluate the effect of direct and indirect pick up of the locator retentive caps and compare the clinical results with those of the manufacturer retentive force.

DETAILED DESCRIPTION:
Patient selection:

For this study, 30 patients were selected from the clinic of Prosthodontic Department, Faculty of Dentistry, Mansoura University.

According to pick up technique for the locator retentive caps, the overdentures will be classified into two groups as follows; Group1: The retentive caps will be picked up by indirect method on the cast then by the direct method Group2: The retentive caps will be picked up in the patient by the direct method first then by the indirect method.

For both groups, the clinical retention will be measured after using pink and blue retentive inserts respectively.

All implants were inserted using computer-guided implant surgery and conventional loading protocol was used.

Evaluation methods The clinical retention of each insert will be calibrated as regards the manufacturer's value.

Also, the laboratory retention will be assessed for the two groups and calibrated as regards the manufacturer's value.

Measurements will be done immediately, three and six months after each overdenture insertion.

ELIGIBILITY:
Inclusion Criteria:

* ● Free from any systemic disease that may interfere with the osseointegration of implants.

  * Patients will have completely edentulous maxilla and mandible for at least 6 months after the last extraction.
  * Patients will have normal maxilla mandibular relationships.
  * Mandibular arch with residual alveolar ridges covered with firmly attached mucosa.
  * The width of the mandibular ridge in the canine area will be sufficient for the installation of the implants in parallel anteroposterior and mesiodistal directions.

Exclusion Criteria:

* medically compromised patients smokers uncontrolled metabolic diseases ( diabetes mellitus ) uncooperative patients

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-08-07 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
measurement of overdenture retention | three months
  measuring the clinical retention of the locator retained mandibular overdenture by forcemeter

SECONDARY OUTCOMES:
marginal bone loss | one year
  measuring crestal bone loss around dental implants in mm by digital radiography
plaque index | one year
  measuring plaque around dental implants using scoring system: score 0; absence plaque , score 1; plaque only detected by a probe passing through the smooth marginal surface of the implant, score 2; plaque can be recognized by naked eye, and score 3; plenty of soft matter.
gingival index | one year
  measuring gingival bleeding using scoring system: 0; no bleeding when a periodontal probe is passed along the mucosal margin, 1;isolated bleeding spots visible, 2; blood forms a confluent red line on the mucosal margin, 3;heavy or profuse bleeding
pocket depth | one year
  measuring pocket depth around dental implants in mm using periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- Christine Ibrahim, Al Mansurah, Egypt